CLINICAL TRIAL: NCT01255618
Title: The Measurement Of Cerebral Oxygenisation With NIRS Method İn Polycythaemic Infants Might Add A Criterion To Indicate PPET?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Zekai Tahir Burak Maternity Teaching Hospital, Zekai Tahir Burak Maternity Teaching Hospital
Other Study IDs: 2
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-11

CONDITIONS: Cerebral Oxygenation; Peripheric Oxygenation; Polycythaemic Infants

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- study group, control group
  Interventions: Device: INVOS 5100

INTERVENTIONS:
Device: INVOS 5100 — Near-infrared range and has been used in newborn infants since 1985. Fibre-optic bundles or optodes are placed either on opposite sides of the tissue being interrogated (usually a limb or the head of a young baby) to measure transmitted light, or close together to measure reflected light. Light enters through one optode and a fraction of the photons is captured by a second optode and conveyed to the measuring device. NIRS uses a frequency band between 650 nm and 1000 nm and relies on three important phenomena: (1) human tissue is relatively transparent to light in the near-infrared region of the spectrum; (2) pigmented compounds known as chromophores absorb light as it passes through biological tissue; and (3) human tissues contain substances whose absorption spectra at near-infrared wavelengths are well defined and depend on their oxygenation status.

SUMMARY:
Near infrared spectrophotometry (NIRS) offers the possibility of noninvasive and continuous bedside investigation of cerebral , renal, mesenteric and peripheric oxygenation and hemodynamics, and changes in newborn period.The aim of the present study is to investigate cerebral oxygenation with NIRS method in polycythaemic infants who underwent partial exchange transfusion.

ELIGIBILITY:
Inclusion Criteria:

term (≥37wk) infants whom determined ≥ 65% haematocrit(Hct) levels

Exclusion Criteria:

Infants with severe congenital malformation, sepsis, intracranial hemorrhage, birth asphyxia were excluded from the study.

Ages: 4 Hours to 48 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm infants who admitted to neonatal intensive care unit.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-11; Primary Completion 2010-12 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
cerebral oxygenation measurement | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zekai Tahir Maternity Teaching Hospital, Ankara, Altındag, Turkey (Türkiye)